CLINICAL TRIAL: NCT00783328
Title: A Clinical Phase 1 Safety And Pharmacokinetic/Pharmacodynamic Study Of PF-00299804 In Patients In Japan With Advanced Malignant Solid Tumors
Brief Title: A Study Of PF-00299804 In Patients In Japan With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A7471005
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasms
Keywords: solid tumor
MeSH Terms: conditions — Neoplasms | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Open label single arm trial
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — Dosage form: 5 mg and 20 mg tablet Dosage: 15 mg, 30 mg and 45 mg, orally, once daily Number of Cycles: until progression or unacceptable toxicity develops.

SUMMARY:
To evaluate safety and tolerability of PF-00299804 in Japanese patients with advanced malignant solid tumors at doses up to the clinically recommended phase 2 dose in non-Japanese studies.

ELIGIBILITY:
Inclusion Criteria:

* Malignant solid tumor with no currently approved treatment
* Adequate functions Bone Marrow, Renal, Liver and Cardiac

Exclusion Criteria:

* Any surgery, radiotherapy within 4 weeks of baseline disease assessments
* Clinically significant abnormalities of the cornea
* Patients with symptomatic brain/central nerve system metastases
* Any clinically significant gastrointestinal abnormalities
* Uncontrolled or significant cardiovascular disease
* Patients with significant interstitial pneumonia or pulmonary fibrosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall safety: type, grade and frequency of all adverse events and laboratory abnormalities | End of study

SECONDARY OUTCOMES:
To explore PD markers | End of study
To evaluate the plasma pharmacokinetics of PF-00299804 in Japanese patients following single and multiple dosing | End of study
To assess any clinical evidence of anti-tumor activity of PF-00299804 per RECIST | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Sunto-gun, Shizuoka, Japan

REFERENCES:
- [Derived] Takahashi T, Boku N, Murakami H, Naito T, Tsuya A, Nakamura Y, Ono A, Machida N, Yamazaki K, Watanabe J, Ruiz-Garcia A, Imai K, Ohki E, Yamamoto N. Phase I and pharmacokinetic study of dacomitinib (PF-00299804), an oral irreversible, small molecule inhibitor of human epidermal growth factor receptor-1, -2, and -4 tyrosine kinases, in Japanese patients with advanced solid tumors. Invest New Drugs. 2012 Dec;30(6):2352-63. doi: 10.1007/s10637-011-9789-z. Epub 2012 Jan 17. PMID 22249430
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471005&StudyName=A%20Study%20Of%20PF-00299804%20In%20Patients%20In%20Japan%20With%20Advanced%20Malignant%20Solid%20Tumors